CLINICAL TRIAL: NCT02673021
Title: MARK 1A Series: Percutaneous Microwave Ablation for Patients With Lung Tumor(s)
Acronym: MARK 1A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding suspended prior to completing enrollment of all participants.
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Shanda Blackmon, M.D., M.P.H., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001758; NCI-2022-10762 (Other: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2016-01-29; First posted 2016-02-03 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Lung Neoplasms; Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Metastatic Cancer to the Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Microwave Ablation (Experimental): Microwave Ablation
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — Microwave tumor ablation is a procedure that uses heat made by an electric current to destroy a tumor (ablation). With imaging equipment, such as ultrasound or CT (computed tomography), and a small incision made in the skin, the tumor is located and treated with radiofrequency energy. The cells that are killed by the microwave ablation are typically not removed but are eventually replaced by fibrosis and scar tissue.

SUMMARY:
Does lung ablation improve clinical outcomes for patients deemed to be surgically high-risk?

DETAILED DESCRIPTION:
Surgical resection is the gold standard treatment for localized non-small cell lung cancer (NSCLC). However, surgery is invasive and not all patients are surgical candidates, thus providing an opportunity for percutaneous microwave ablation, for both primary and metastatic disease. Patients that are deemed inoperable are typically treated with other targeted therapies such as radiofrequency ablation (RFA), cryoablation and stereotactic body radiation therapy (SBRT), or systemic therapies. Percutaneous microwave ablation (MWA) is an alternative option for targeted treatment of cancer. Microwave tumor ablation is a procedure that uses heat made by an electric current to destroy a tumor (ablation). With imaging equipment, such as ultrasound or CT (computed tomography), and a small incision made in the skin, the tumor is located and treated with radiofrequency energy. The cells that are killed by the microwave ablation are typically not removed but are eventually replaced by fibrosis and scar tissue. Patients will be followed for 1 year by contrast enhanced chest CT, chest PET/CT and chest PET/MRI to evaluate lesion outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years old.
* Subject is able to understand the study procedures and provide informed consent.
* Subject is willing and able to complete the entire study as specified in the protocol, including the follow-up visits.
* Subject has lung lesion that is biopsy-proven cancer (of any type) or suspicious, with confirmation at the time of the procedure.
* Lung lesion(s) are reachable/treatable per clinician opinion.
* Subject can have other location of disease if it is controlled, or there are plans for control.
* Subject has 1 or more lung nodules (not more than 10), that have a mean diameter <3 cm on axial CT scan.
* Life expectancy ≥6 months

Exclusion Criteria:

* Subject is pregnant or breast feeding.
* Subject has a significant clinical disease or condition, e.g. cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematological, psychiatric or neurologic that would preclude enrollment, as determined by the primary investigator.
* Subject has another location of disease that is not controlled, and there are no plans for control.
* Subject has more than 10 lung nodules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Efficacy of microwave ablation. | 3 months
  Efficacy is defined as achieving the technical success = complete ablation = achieving ablation zone size predicted/necessary for treatment.
Assessment of patient adverse events as defined by CTCAE. | 3 months
  The safety evaluation is based on the major complication rates of performing microwave ablation. The intent is to determine if the results are within acceptable range of what is reported for RFA, cryoablation and surgery. If the microwave ablation has a safety profile that is outside the "standard of care" range, then the procedure would be deemed unacceptable and no further studies of the current generation of microwave ablation would be recommended. The study team has deemed major complication rates of 50% or greater as outside of the "standard of care" range.

SECONDARY OUTCOMES:
Pathological response in patients receiving microwave ablation. | 1 year
  Clinical samples and imaging will be examined to determine pathological response.

CONTACTS AND LOCATIONS:
Overall Officials: Shanda Blackmon, MD, MPH, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials